CLINICAL TRIAL: NCT02245880
Title: A Comparison of Glidescope and ILMA in Simulated Sercial Spine Injury
Brief Title: Tracheal Intubation With Collar Immobilisation : a Comparison of Glidescope and Fastrach
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Zehra Ipek ARSLAN, Assistant Professor, Kocaeli University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: KOÜ KAEK 2013/33
Record Dates: First submitted 2014-04-17; First posted 2014-09-22 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2015-03

CONDITIONS: Injury of Cervical Spine
Keywords: cervical spine; intubating laryngeal mask airway; Glidescope videolaryngoscope; collar

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Glidescope videolaryngoscope (Active Comparator): cervical collar was applied to 47 patients then facemask ventilations were recoded intubated with Glidescope and insertion time: handling of the device till the good glottic visualisation intubation time: handling of the device till the capnography appears mucosal damage: bloodstain on the device after removal heart rate preinduction heart rate postinduction heart rate postinsertion heart rate postintubation mean arterial pressure preinduction mean arterial pressure postinduction mean arterial pressure postinsertion mean arterial pressure postintubation wrere recorded. postoperative minor complications were recorded.
  Interventions: Device: Glidescope
- Intubating laryngeal mask airway (Active Comparator): cervical collar was applied to 47 patients then facemask ventilations through the collar were recorded and intubated with ILMA insertion time: handling of the device till the good glottic visualisation appears intubation time: handling of the device till the capnography appears mucosal damage: bloodstain on the device heart rate preinduction heart rate postinduction heart rate posinsertion heart rate postintubation mean arterial pressure preinduction mean arterial pressure postinduction mean arterial pressure postinsertion mean arterial pressure postintubation
  Interventions: Device: ILMA

INTERVENTIONS:
Device: Glidescope — videolaryngoscope
  Arms: Glidescope videolaryngoscope
Device: ILMA — handling of the device till the optimal ventilation achieved
  Other Names: FASTRACH
  Arms: Intubating laryngeal mask airway

SUMMARY:
Intubation must be done with utmost care in cervical trauma patients. cervical spine motion must be minimized and intubation must be fast. The aim of this study was to compare the effectiveness of fastrach and glidescope. 18-65 years of age , ASA I-II 100 patients undergoing elective surgery were enrolled in this trial. After standard monitorisation including EKG , noninvasive blood pressure, pulse oximetry, anesthesia was induced with propofol and fentanyl. rocuronium was then administered for muscle relaxation. Patients were divided into two groups glidescope and fastrach. Rigid collar was placed then patients were intubated with one of these devices. Mask ventilations with or without collar were recorded. insertion times, intubation times of the devices were recorded. Peroperative hemodynamic parameters and postoperative minor complications were also recoded.

DETAILED DESCRIPTION:
inclusion criteria: ASA I-II , 18-60 years of age undergoing elective surgery requiring intubation exclusion criteria:

- pregnancy reflux nonfasted head and neck tumors recent flue in 2 weeks

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age
* ASA I-II
* requiring intubation
* BMI<35

Exclusion Criteria:

* less than 18 or higher than 65
* ASA III-IV
* BMI> 35
* PREGNANT
* head and neck tumors

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2014-04; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
intubation times | From handling of the device till intıbation

SECONDARY OUTCOMES:
Heart rate | From Preoperative heart rate till 15 minutes After intubation
Mean arterial pressure | From preinduction till 15 minutes after intubation

OTHER OUTCOMES:
minor complications | From the end of surgery till 2 hours postoperatively
Mucosal damage | Bloodstain on the device after removal

CONTACTS AND LOCATIONS:
Overall Officials: Zehra I ARSLAN, Specialist, Principal Investigator — Anesthesiology and Reanimation
Locations (1):
- Kocaeli University School of Medicine, Kocaeli, Turkey (Türkiye)